CLINICAL TRIAL: NCT05028283
Title: Autologous Fat Cells Transfer for the Treatment of Atrophic Post Acne Scars: Clinical Trail
Brief Title: Treatment of Atrophic Post Acne Scars by Fat Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDMS-Derma-01-2021
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Atrophic Acne Scars
Keywords: Acne- atrophic scars - autologous fat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): patients with atrophic acne scars on the cheeks who will reviewing the dermatological clinics at the Dermatology and Venereology Hospital at least 69 patients they will be undergo fat grafting for one session and will be follow up for 6 months after the procedure
  Interventions: Procedure: Fat Grafting

INTERVENTIONS:
Procedure: Fat Grafting — This single-center, clinical trial will assess the efficacy and tolerability of the autologous fat grafting when used on men and women with atrophic acne scars on the cheeks

SUMMARY:
This single-center, clinical trial consists of a one autologous fat grafting treatment followed by1-week , 1month , 3-month and 6-month post-treatment visits in order to assess the efficacy and complications of fat grafting when used for facial atrophic acne scars on cheeks.

DETAILED DESCRIPTION:
This investigation, pilot study will evaluate the safety and efficacy of autologous fat grafting for the treatment of atrophic acne scarring on cheeks. Overall assessment of clinical outcome and safety will be based clinic visits and evaluation of pre- and post- procedural on the Goodman-Barron scale.

The subject's assessment of satisfaction will be characterized using a non-parametric assessment scale at the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophic post acne scars on the cheeks, between 20 - 40 years old
* Not to apply other treatments a month before the procedure
* Informed consent to enter the study

Exclusion Criteria:

* First grade of Goodman - Barron scale.
* A systemic or associated skin disease that may affect the results of the study
* patients with chronic consumption of nonsteroidal anti-inflammatory drugs (NSAIDs) or other non-aggregating agents.
* Patients with acne in the acute stage
* Pregnancy and breastfeeding
* Tendency to form keloids

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
• Change in atrophic acne scars assessment | Baseline and 6 Months
  Acne scars will be used to evaluate efficacy of treatment using the Goodman- Barron scale [which is an acne scars severity scale divided into 4 grades
  * First grade consists of hyper-or hypopigmented flat marks
  * Second grade consists of mild atrophy or hypertrophy that may not be obvious at social distances of 50 cm or greater and may be covered adequately by makeup
  * Third grade consists of moderate atrophic or hypertrophic scarring that is obvious at social distances of 50 cm or greater and is not covered easily by makeup or the normal shadow
  * Fourth grade severe atrophic or hypertrophic scarring that is obvious at social distances of 50 cm or greater and is not covered easily by makeup or the normal shadow].
  The grade of acne scars from final visit will be compared to their baseline grade visually evaluated by the study team.
Change in patient satisfaction | 3 Months, and 6 Months
  The modified global aesthetic improvement scale for patient evaluation module which consists of 5 degrees
  * Exceptionally improved [The ideal result has been achieve]
  * much improved[The result is much improved but suboptimal]
  * Improved[The result is improved but an additional procedure is recommended ]
  * no difference[The result is the same when compared with the preoperative state]
  * Worse[The result is worse when compared with the preoperative state] This module will be administered 3monts and 6 months postoperatively to analyze satisfaction and aesthetic perception of the result.

SECONDARY OUTCOMES:
Change in Infection existence | 1 week, 1 month, 3 months and 6 Months
  Patients will be examined after procedure to check existence of infection and will be monitored until it will heal.
Change in Bruising Status | Baseline ,1 week 1 month,3 months and 6 Months
  Patients will be examined after procedure to check bruising status and will be monitored until it will disappear
Change in Erythema Presence | Baseline ,1 week ,1 month,3 months and 6 Months
  Patients will be examined after procedure to check erythema presence and will be monitored until it will disappear
Change in Swelling Status | Baseline ,1 week 1month,3 months and 6 Months
  Patients will be examined after procedure to check swelling status and will be monitored until it will disappear
Change in Irregularity Presence | Baseline and 6 Months
  Patients will be examined after procedure to check irregularity presence at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Rahaf Alkhouli, MSc, Principal Investigator — Dermatology Department, University of Damascus Medical School
Locations (1):
- Dermatology and Venereology Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams HC, Dellavalle RP, Garner S. Acne vulgaris. Lancet. 2012 Jan 28;379(9813):361-72. doi: 10.1016/S0140-6736(11)60321-8. Epub 2011 Aug 29. PMID 21880356
- [Background] Goulden V, McGeown CH, Cunliffe WJ. The familial risk of adult acne: a comparison between first-degree relatives of affected and unaffected individuals. Br J Dermatol. 1999 Aug;141(2):297-300. doi: 10.1046/j.1365-2133.1999.02979.x. PMID 10468803
- [Background] Boen M, Jacob C. A Review and Update of Treatment Options Using the Acne Scar Classification System. Dermatol Surg. 2019 Mar;45(3):411-422. doi: 10.1097/DSS.0000000000001765. PMID 30856634
- [Background] Thiboutot D, Gollnick H, Bettoli V, Dreno B, Kang S, Leyden JJ, Shalita AR, Lozada VT, Berson D, Finlay A, Goh CL, Herane MI, Kaminsky A, Kubba R, Layton A, Miyachi Y, Perez M, Martin JP, Ramos-E-Silva M, See JA, Shear N, Wolf J Jr; Global Alliance to Improve Outcomes in Acne. New insights into the management of acne: an update from the Global Alliance to Improve Outcomes in Acne group. J Am Acad Dermatol. 2009 May;60(5 Suppl):S1-50. doi: 10.1016/j.jaad.2009.01.019. PMID 19376456
- [Background] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456
- [Background] Coleman SR. Facial augmentation with structural fat grafting. Clin Plast Surg. 2006 Oct;33(4):567-77. doi: 10.1016/j.cps.2006.09.002. PMID 17085224
- [Background] Zeltzer AA, Tonnard PL, Verpaele AM. Sharp-needle intradermal fat grafting (SNIF). Aesthet Surg J. 2012 Jul;32(5):554-61. doi: 10.1177/1090820X12445082. PMID 22745443
- [Background] Lindenblatt N, van Hulle A, Verpaele AM, Tonnard PL. The Role of Microfat Grafting in Facial Contouring. Aesthet Surg J. 2015 Sep;35(7):763-71. doi: 10.1093/asj/sjv083. Epub 2015 Jun 2. PMID 26038369
- [Background] Tonnard P, Verpaele A, Peeters G, Hamdi M, Cornelissen M, Declercq H. Nanofat grafting: basic research and clinical applications. Plast Reconstr Surg. 2013 Oct;132(4):1017-1026. doi: 10.1097/PRS.0b013e31829fe1b0. PMID 23783059
- [Background] Goodman GJ, Baron JA. Postacne scarring: a qualitative global scarring grading system. Dermatol Surg. 2006 Dec;32(12):1458-66. doi: 10.1111/j.1524-4725.2006.32354.x. PMID 17199653
- [Background] Sezgin B, Ozmen S. Fat grafting to the face with adjunctive microneedling: a simple technique with high patient satisfaction. Turk J Med Sci. 2018 Jun 14;48(3):592-601. doi: 10.3906/sag-1711-42. PMID 29914257